CLINICAL TRIAL: NCT07253636
Title: An Examination of the Effects of the Social and Emotional Development Support Program on Adolescents' Sense of Belonging, Meaning in Life, Emotional Authenticity, Well-Being, and Psychological Resilience
Brief Title: Social and Emotional Development Support Program for Adolescents: Effects on Belonging, Meaning in Life, Authenticity, Well-Being, and Resilience
Acronym: SEDESP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Didem Aslanyürek, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DIDEM-ASLANYUREK-INTERV-2025; E-68552689-302.08-00003594733 (Other: Hacettepe University Social and Human Sciences Research Ethics Committee)
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Adolescent Social and Emotional Development
Keywords: Adolescents; Social and emotional development; Well-being; Belonging; Meaning in life; Emotional authenticity; Resilience

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the experimental and control groups before baseline measurements. After the groups are determined, pre-test data will be collected from both groups. The Social and Emotional Developmental Support Program will be administered to the experimental group, while the control group will receive no intervention during the study period. Following the completion of the program, post-test data will be collected from both groups to evaluate the effectiveness of the intervention.
Who Masked: Participant
Masking Description: Participants were not informed whether their school was assigned to the intervention or control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social and Emotional Developmental Support Program (Experimental): Participants in this group will receive the Social and Emotional Developmental Support Program, which aims to enhance adolescents' sense of belonging, meaning in life, emotional authenticity, well-being, and resilience. The program will be implemented over several structured sessions conducted in a school setting.
  Interventions: Behavioral: Social and Emotional Developmental Support Program
- No Intervention (Assessment Only Control Group) (No Intervention): Participants in this group will not receive any intervention during the study period. They will complete the same pre- and post-test assessments as the experimental group.

INTERVENTIONS:
Behavioral: Social and Emotional Developmental Support Program — A structured program designed to promote adolescents' social and emotional development. The program includes interactive sessions aimed at enhancing belonging, meaning in life, emotional authenticity, well-being, and resilience. It will be implemented in a school setting through group-based activities and reflective discussions.
  Arms: Social and Emotional Developmental Support Program

SUMMARY:
This study aims to examine the effectiveness of the Social and Emotional Developmental Support Program on adolescents' sense of belonging, meaning in life, emotional authenticity, well-being, and resilience. The study will be conducted with 9th-grade students studying in Defne district of Hatay, Türkiye, one of the regions affected by the Kahramanmaraş-centered earthquake that occurred on February 6, 2023. A pre-test/post-test control group experimental design will be used to evaluate the effectiveness of the program.

DETAILED DESCRIPTION:
This study aims to examine the effects of the Social and Emotional Developmental Support Program, which will be implemented with ninth-grade students studying in the Defne district of Hatay, on adolescents' sense of belonging, meaning in life, emotional authenticity, well-being, and resilience. The research will be carried out with adolescents living in Defne, one of the districts of Hatay most affected by the Kahramanmaraş-centered earthquake that occurred in Türkiye on February 6, 2023. The study is designed as a pre-test/post-test control group experimental design. Participants will be randomly assigned to experimental and control groups. The experimental group will receive the Social and Emotional Developmental Support Program, whereas no intervention will be provided to the control group during the study period. Data will be collected using a demographic information form and standardized instruments assessing adolescents' sense of belonging, meaning in life, emotional authenticity, well-being, and resilience. The findings are expected to contribute to the social and emotional development of adolescents affected by the earthquake and to enrich the existing body of literature.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged between 14 and 15 years
* Ninth-grade students enrolled in public high schools located in the Defne district of Hatay
* Individuals who resided in the Defne district on February 6, 2023
* Students who voluntarily agree to participate and whose parental consent has been obtained
* Students who are able to attend all program sessions regularly

Exclusion Criteria:

* Students who did not reside in the Defne district on February 6, 2023
* Students with special educational needs or those reported by school counselors or parents to have developmental or psychiatric diagnoses
* Students who are simultaneously participating in another psychosocial intervention program
* Students with cognitive limitations that prevent them from completing the study assessments

Ages: 14 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2025-12-26 (Estimated)

PRIMARY OUTCOMES:
The General Belongingness Scale | Baseline (pre-test) and after completion of the intervention (approximately 11 weeks).
  Participants' sense of belonging will be assessed using the General Belongingness Scale. The General Belongingness Scale is answered on a four-point Likert scale with the options "(1) Strongly disagree, (2) Somewhat disagree, (3) Mostly agree, (4) Strongly agree." Six items represent the rejection/exclusion dimension, while the remaining six items reflect the acceptance/inclusion dimension. When all 12 items are evaluated together, a total belongingness score is obtained. In this context, higher total scores indicate higher levels of general belongingness among adolescents.
Meaning in Life Questionnaire | Baseline (pre-test) and after completion of the intervention (approximately 11 weeks).
  Participants' perceived meaning in life will be assessed using the Meaning in Life Questionnaire. Higher scores on the Presence of Meaning subscale indicate that individuals perceive their lives as more meaningful and purposeful, whereas higher scores on the Search for Meaning subscale reflect greater efforts to find or develop meaning in life. When calculating the total score by reverse-coding the Search subscale, a higher overall score signifies a stronger sense of meaning in life.
Emotional Authenticity Scale | Baseline (pre-test) and after completion of the intervention (approximately 11 weeks).
  Participants' emotional authenticity will be measured using the Emotional Authenticity Scale. The Emotional Authenticity Scale is a 20-item self-report measure assessing the extent to which individuals express their emotions in a genuine, coherent, and self-consistent manner. Items are rated on a 1-5 Likert scale. Five items from the "Acceptance of External Influence" subscale and seven items from the "Emotional Avoidance" subscale are reverse-scored. Higher total scores indicate greater emotional authenticity.
EPOCH Well-being Scale | Baseline (pre-test) and after completion of the intervention (approximately 11 weeks).
  Participants' well-being levels will be assessed using the EPOCH Well-Being Measure. The scale consists of five subscales and a total of 20 items. Higher scores on each subscale indicate a greater level of the specific characteristic assessed by that dimension. In addition, the scale provides an overall well-being score. During scoring, mean scores are calculated for each subscale as well as for the total scale.
Psychological Resilience Attitude and Skills Scale | Baseline (pre-test) and after completion of the intervention (approximately 11 weeks).
  Participants' resilience levels will be measured using the Resilience Attitude and Skill Scale. It is a 34-item, single-factor measurement tool rated on a four-point Likert scale. There are no reverse-scored items in the scale. Higher scores indicate higher levels of psychological resilience.

CONTACTS AND LOCATIONS:
Locations (1):
- Defne Public High Schools, Hatay, Defne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared due to ethical considerations and confidentiality requirements. The dataset includes sensitive information from adolescent participants collected in a school setting, and sharing such data could compromise participant privacy. The data will not be shared with third parties except for scientific purposes within the approved research framework.